CLINICAL TRIAL: NCT05329038
Title: Immunogenicity，Safety and Cross - Immune Response With Mutant Strains of the Third Dose Using Inactivated COVID-19 Vaccine in Population Aged 18 Years and Above
Brief Title: Immunogenicity，Safety and Cross - Immune Response With Mutant Strains of a Third Dose of an Inactivated COVID-19 Vaccine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sinovac Life Sciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-nCOV-MA4009-SD
Record Dates: First submitted 2022-04-12; First posted 2022-04-14 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — sinovac COVID-19 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adult group (Experimental): 90 subjects aged 18-59 years received two dose inactivated COVID-19 vaccine in primary immunization will receive the booster immunization (the third dose )of inactivated COVID-19 vaccine.
  Interventions: Biological: Inactivated COVID-19 Vaccine
- Elderly group (Experimental): 90 elderly aged 60 year and older received two dose inactivated COVID-19 vaccine in primary immunization will receive the booster immunization (the third dose )of inactivated COVID-19 vaccine.
  Interventions: Biological: Inactivated COVID-19 Vaccine

INTERVENTIONS:
Biological: Inactivated COVID-19 Vaccine — 600SU inactivated virus in 0·5 mL of aluminium hydroxide solution per injection
  Other Names: CoronaVac

SUMMARY:
This is a phase Ⅳ follow-up clinical trial based on the previous Phase Ⅳ clinical trial of an inactivated COVID-19 vaccine (CoronaVac) manufactured by Sinovac Life Sciences Co., Ltd.The purpose of this study is to evaluate the immunogenicity,safety and cross-immune response of booster immunization using COVID-19 vaccine,to compare the similarities and differences of immune responses between primary immunization and booster immunization and to detect antibody against hepatitis A and evaluate the immune persistence of the one dose immunization schedule of hepatitis A vaccine in healthy population aged 18 years and older.

DETAILED DESCRIPTION:
This study is a phase 4 clinical trial to evaluate the immunogenicity,safety and cross-immune response of booster immunization using COVID-19 vaccine，to compare the similarities and differences of immune responses between primary immunization and booster immunization and to detect antibody against hepatitis A and evaluate the immune persistence of the one dose immunization schedule of hepatitis A vaccine in healthy population aged 18 years and older. The experimental vaccine is manufactured by Sinovac Life Sciences Co., Ltd.. A total of 180 healthy subjects received two dose of inactivated COVID-19 vaccine (CoronaVac) based on primary immunization in previous Phase Ⅳ clinical trial will be enrolled, including 90 adults aged 18-59 years and 90 elderly elderly aged 60 years and older.Subjects in each age group will receive the booster immunization of CoronaVac(the third dose) and will be collected blood sample before booster immunization and 14 days after booster immunization.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the clinical studies on the safety and immunogenicity of Inactivated COVID-19 Vaccine combined immunization with 23-valent pneumococcal polysaccharide vaccine in Rushan city, Shandong Province from July to October 2021;
* The interval between complete immunization with two doses of COVID-19 vaccine is 6-8 months;
* Subjects will be willing to participate in the study and follow the study procedure to collect venous blood;
* Proven legal identity;

Exclusion Criteria:

* History of asthma, history of allergy to the vaccine or vaccine components,or serious adverse reactions to the vaccine, such as urticaria, dyspnea,and angioedema;
* Severe neurological disease (epilepsy, convulsions or convulsions) or mental illness;
* Fever at the time of vaccination, or acute onset of chronic disease, or uncontrolled severe chronic disease, or acute disease;
* Pregnancy or lactation;
* Receipt of attenuated live vaccines in the past 14 days;
* Receipt of inactivated or subunit vaccines in the past 7 days
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2022-06-19 (Actual); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rate of neutralizing antibody against Prototype SARS-CoV-2 | 14 days after the booster immunization of inactivated COVID-19 vaccine
  The seroconversion rate of neutralizing antibody against Prototype SARS-CoV-2 at 14 days after the booster immunization of inactivated COVID-19 vaccine.

SECONDARY OUTCOMES:
Seropositive rate of neutralizing antibody against Prototype SARS-CoV-2 | 14 days after the booster immunization of inactivated COVID-19 vaccine
  The seropositive rate of neutralizing antibody against Prototype SARS-CoV-2 at 14 days after the booster immunization of inactivated COVID-19 vaccine.
GMT of neutralizing antibody against Prototype SARS-CoV-2 | 14 days after the booster immunization of inactivated COVID-19 vaccine
  The GMT of neutralizing antibody against Prototype SARS-CoV-2 at 14 days after the booster immunization of inactivated COVID-19 vaccine.
GMI of neutralizing antibody against Prototype SARS-CoV-2 | 14 days after the booster immunization of inactivated COVID-19 vaccine
  The GMI of neutralizing antibody against Prototype SARS-CoV-2 at 14 days after the booster immunization of inactivated COVID-19 vaccine.
Seroconversion rate of neutralizing antibody against SARS-CoV-2 strains | 14 days after the booster immunization of inactivated COVID-19 vaccine
  The seroconversion rate of neutralizing antibody against SARS-CoV-2 strains at 14 days after the booster immunization of inactivated COVID-19 vaccine.
Seropositive rate of neutralizing antibody against SARS-CoV-2 strains | 14 days after the booster immunization of inactivated COVID-19 vaccine
  The seropositive rate of neutralizing antibody against SARS-CoV-2 strains at 14 days after the booster immunization of inactivated COVID-19 vaccine.
GMI of neutralizing antibody against SARS-CoV-2 strains | 14 days after the booster immunization of inactivated COVID-19 vaccine
  The GMI of neutralizing antibody against SARS-CoV-2 strains at 14 days after the booster immunization of inactivated COVID-19 vaccine.
GMT of neutralizing antibody against SARS-CoV-2 strains | 14 days after the booster immunization of inactivated COVID-19 vaccine
  The GMT of neutralizing antibody against SARS-CoV-2 strains at 14 days after the booster immunization of inactivated COVID-19 vaccine.
Seropositive rate of antibody against hepatitis A | 6-8 months after vaccination of Hepatitis A vaccine
  Seropositive rate of antibody against hepatitis A 6-8 months after vaccination of Hepatitis A vaccine.
GMC of antibody against hepatitis A | 6-8 months after vaccination of Hepatitis A vaccine
  GMC of antibody against hepatitis A 6-8 months after vaccination of Hepatitis A vaccine.
Incidence rate of adverse reactions | 0-28 days after booster immunization with COVID-19 vaccine.
  Incidence rate of adverse reactions within 0-28 days after booster immunization with COVID-19 vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Master, Principal Investigator — Shandong Provincial Center for Disease Control and Prevention
Locations (1):
- Rushan City Center for Disease Control and Prevention, Weihai, Shandong, China